CLINICAL TRIAL: NCT00802633
Title: Radical Cystectomy: Can We Improve Our Surgical Technique With the Ligasure Impact Tissue-Sealing Device?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment was stopped after eighty patients were enrolled.
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, SChang, MD, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 081018
Record Dates: First submitted 2008-12-03; First posted 2008-12-05 (Estimated); Results first posted 2014-02-11 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2013-12

CONDITIONS: Bladder Cancer; Hemostasis
Keywords: Tissue sealing device; Articulating stapling device; Radical cystectomy
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stapling device (Active Comparator): Efficacy of stapling device during radical cystectomy
  Interventions: Device: Stapling device during radical cystectomy
- Ligasure Device (Active Comparator): Efficacy of ligasure tissue sealing device during radical cystectomy
  Interventions: Device: Ligasure tissue sealing device

INTERVENTIONS:
Device: Stapling device during radical cystectomy — Hemostasis
  Other Names: Ethicon articulating stapler
  Arms: Stapling device
Device: Ligasure tissue sealing device — Efficacy of tissue sealing device during hemostasis
  Other Names: Tissue sealing device
  Arms: Ligasure Device

SUMMARY:
Evaluate the utility/safety of an FDA-approved tissue sealing device during radical cystectomy as compared to an FDA-approved stapling device.

ELIGIBILITY:
Inclusion Criteria:

* Muscle invasive bladder cancer
* Male/Female gender

Exclusion Criteria:

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-11; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sam S Chang, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stapling Device | Ligasure Device
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stapling Device | Ligasure Device | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (9.6) | 68.5 (7.9) | 67.15 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 37 | 33 | 70
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Estimated Blood Loss
Time Frame: Perioperative
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Stapling Device | Ligasure Device
Number analyzed (Participants) | 40 | 40
milliliters | 686.5 (406.1) | 707.5 (570.8)

2. Secondary Outcome: Operating Room Time in Minutes
Time Frame: Intraoperative time
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Stapling Device | Ligasure Device
Number analyzed (Participants) | 40 | 40
minutes | 262.1 (74.9) | 272.9 (73.3)

ADVERSE EVENTS:
Arm/Group | Stapling Device | Ligasure Device
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

LIMITATIONS AND CAVEATS:
Study terminated after 80 subjects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No